CLINICAL TRIAL: NCT06549244
Title: A Pilot Study on Inspiratory Dynamics and the Effect of Body Mass Index on Respiratory Outcomes After Temporary Hemi Diaphragmatic Paresis Related to Brachial Plexus Blocks
Brief Title: Preoperative Maximum Inspiratory Pressure and Outcomes After Interscalene Block in Obese Patients
Status: Completed | Type: Observational
Sponsor: University of North Carolina, Chapel Hill (Other)
Responsible Party: Sponsor
Other Study IDs: 23-0924
Record Dates: First submitted 2024-07-31; First posted 2024-08-12 (Actual); Last update posted 2024-08-12 (Actual); Status verified 2024-07

CONDITIONS: Dyspnea After Interscalene Nerve Block

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Block, Non-obese: Non-obese, Body Mass Index (BMI)<30, receiving interscalene block and general anesthesia for shoulder surgery
  Interventions: Diagnostic Test: Maximum Inspiratory Pressure monitoring
- Block, Obese: Class 2 or higher Obese, BMI>35, receiving interscalene block and general anesthesia for shoulder surgery
  Interventions: Diagnostic Test: Maximum Inspiratory Pressure monitoring
- Control: control group, included non-shoulder surgery patients receiving general anesthesia only
  Interventions: Diagnostic Test: Maximum Inspiratory Pressure monitoring

INTERVENTIONS:
Diagnostic Test: Maximum Inspiratory Pressure monitoring — Lung volumes, pressures and breathlessness scores to be measured in pre and post operative phase of care on the same day
  Other Names: Spirometry measurements, Modified Borg breathlessness questionnaire

SUMMARY:
The study aims to explore if Maximum Inspiratory Pressure can predict postoperative breathlessness in obese patients receiving interscalene blocks for shoulder surgery.

The main question is: does baseline Maximum Inspiratory Pressure have any association with postoperative breathlessness after interscalene blocks in class 2 or higher obese patients (BMI>35).

Preoperative and postoperative lung volumes, pressures, breathlessness score and respiratory outcomes will be measured on participants already receiving shoulder surgery with interscalene blocks.

ELIGIBILITY:
Inclusion Criteria Groups 1 and 2

* Adults >18 years of age receiving shoulder surgery with preoperative interscalene block and general anesthesia;
* Speak English;

Group 3

· Adults >18 years of age receiving cystoscopy or lower extremity procedures receiving general endotracheal anesthesia

Exclusion Criteria All Groups

* Less than 18 years of age;
* currently pregnant;
* currently incarcerated;
* those with significant neuromuscular disease, tracheo-bronchial structural abnormalities, severe respiratory or severe cardiovascular comorbidity;
* those undergoing intra-abdominal or intrathoracic surgeries due to the potential to independently effect breathing

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients presenting for shoulder surgery with preoperative interscalene block (Groups 1 and 2). Group 3 includes adult patients presenting for non thoracic, non abdominal surgery under general anesthesia.
Sampling Method: Probability Sample
Enrollment: 45 (Actual)
Dates: Start 2023-07-01 (Actual); Primary Completion 2023-11-28 (Actual); Study Completion 2024-01-10 (Actual)

PRIMARY OUTCOMES:
Incidence of Moderate to Severe Breathlessness | Baseline (Arrival to pre-operative phase), Recovery (Immediately post-surgical, up to 3 hours)
  Score of 3 or above on Modified Borg Breathlessness Scale

SECONDARY OUTCOMES:
Oxygen Saturation in post-anesthesia care unit | Recovery (Immediately post-surgical, up to 3 hours)
  Measured by pulse oximetry
Post-anesthesia care unit length-of-stay | Recovery (Immediately post-surgical, up to 3 hours)
  Total time spent in post-operative phase of care
Duration of Oxygen supplementation in post-anesthesia care unit | Recovery (Immediately post-surgical, up to 3 hours)
  Total duration of oxygen supplementation in post-operative phase of care

CONTACTS AND LOCATIONS:
Overall Officials: Monika Nanda, Principal Investigator — University of North Carolina
Locations (1):
- University of North Carolina, Chapel Hill, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No